CLINICAL TRIAL: NCT01771679
Title: A Phase I/II, Open-Label Study to Assess the Safety, Tolerability, and Preliminary Efficacy of a Single Intravenous Dose of Allogeneic Mesenchymal Bone Marrow Cells to Subjects for Cutaneous Photoaging
Brief Title: Safety Study of Bone Marrow Derived Stem Cells on Patients With Cutaneous Photoaging
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Stemedica Cell Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STEM 102-M
Record Dates: First submitted 2013-01-16; First posted 2013-01-18 (Estimated); Last update posted 2022-10-31 (Actual); Status verified 2020-10

CONDITIONS: Chronic Effect of Ultraviolet Radiation on Photoaged Skin; Dermatologic Disorders
Keywords: Mesenchymal Stem Cells; Bone Marrow Cells; Allogeneic Transplantation; Skin Wrinkling; Solar Aging of Skin; Intravenous Administration
MeSH Terms: conditions — Skin Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Allogeneic Mesenchymal Bone Marrow Cells (Experimental): 1550 nm Fraxel laser treatment (6-8 mJ, Level 2) to full face followed by IV infusion of Allogeneic Mesenchymal Bone Marrow Cells (0.5, 1.0, or 1.5 million cells/kg, up to 150 million cells)
  Interventions: Biological: Allogeneic Mesenchymal Bone Marrow Cells

INTERVENTIONS:
Biological: Allogeneic Mesenchymal Bone Marrow Cells — Subjects in Part 1, Cohorts 1-3 will receive a 1550 nm Fraxel laser (6-8 mJ, Level 2) treatment on the face followed by a single intravenous infusion of 0.5, 1.0, or 1.5 million mesenchymal cells per kg of body weight, not to exceed 150 million cells. Subjects in Part 2 will receive a 1550 Fraxel laser (6-8 mJ, Level 2) treatment on the face followed by a single intravenous infusion of mesenchymal cells at the Maximum Tolerated Dose, as determined by the safety results of Part 1. The dose in Part 2 is 1.5 million cells per kg, not to exceed a total of 150 million cells.

SUMMARY:
The purpose of this study is to determine whether a one-time injection of allogeneic mesenchymal bone marrow cells is safe and beneficial in the treatment of photodamage on the face.

DETAILED DESCRIPTION:
Mesenchymal stem cells (MSCs) have been isolated from a number of sources, including bone marrow, adipose tissue, and peripheral blood. The MSCs manufactured for this study are a subset of non-hematopoietic stem cells derived from the bone marrow of healthy, adult donors. These cells have the ability to migrate to areas of injury in the body and can differentiate into multiple cell types, including cutaneous cells. In addition to contributing directly to repair of the skin by replacing damaged cells, MSCs also stimulate the body's own cells to regenerate.

Though an increasing number of patients are seeking remedies for photoaged skin, current treatments, ranging from topical medications to laser peels, are not ideal methods for addressing the medical need. Because MSCs have been shown in clinical and non-clinical applications to be useful in wound healing, it is also possible that the cells will have a similar effect in skin rejuvenation.

In the present study, we will determine the efficacy and safety of intravenously delivered MSCs in otherwise healthy patients with significant cutaneous photodamage.

ELIGIBILITY:
Key Inclusion Criteria:

* Males and Females 40-70 years of age
* Good general health
* Fitzpatrick skin type I-III
* Fitzpatrick Wrinkle Scale class III. Fine to deep wrinkles, numerous lines with or without redundant skin folds
* Ability to understand and provide signed informed consent
* Reasonable expectation that subject will attend all scheduled safety follow-up visits
* Reasonable expectation that subject will maintain skin care regimen for the duration of the trial
* Adequate organ function

Key Exclusion Criteria:

* History of malignant neoplasm within the past 5 years, or Stage 3 or 4 of any cancer at any time
* History of melanoma, leukemia, or lymphoma (any stage)
* Persistent pre-cancerous lesions (e.g., actinic keratosis)
* Active cutaneous infection of the head and/or neck
* Active cutaneous neoplasm in the treatment area
* Topical use of any anti-aging creams on the head and/or neck; if used, subject must agree to discontinue for the one year of follow-up on study
* Cosmetic or surgical treatment on face/neck in 6 months before study (includes laser, chemical peels, fillers, botulinum toxin)
* Prior treatment with stem cells
* Positive for hepatitis B, C or HIV
* Abnormal and clinically significant findings on screening ECG
* Abnormal and clinically significant findings on screening CT scan of the chest (without contrast)
* Clinically significant medical condition for which participation in the study would pose a safety risk to the subject
* Major surgery within 4 weeks of Study Day 1
* Participation in another study with an investigational drug or device within 3 months prior to stem cell administration
* Participation in another study concurrent with the one-year duration of the trial
* History within the past year of drug or alcohol abuse
* Females known to be pregnant, lactating or having a positive pregnancy test (will be tested during screening) or planning to become pregnant during the study
* Sexually active males and females of child-bearing potential must use an effective method of birth control for duration of the study (approximately 13 months from the screening visit)
* Allergies to bovine and porcine products

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2015-07-01 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
MSC Safety and Tolerability | 1 year
  The primary endpoint will be the safety and tolerability of IV administration of allogeneic mesenchymal bone marrow cells (aMBMC) during the twelve month study period as determined by the incidence and severity of adverse events, clinically significant changes on clinical laboratory tests, vital signs, physical and cutaneous examinations, 12 lead ECGs and CT scans of the chest (without contrast)

SECONDARY OUTCOMES:
MSC Efficacy | 12 months
  * VISIA-CR 2D photography
  * PRIMOS 3D images of face and neck
  * VECTRA 3D photography
  * Punch biopsy from the lateral canthal area to examine changes in decorin, fibrillin, elastin, MMPI, and procollagen-1
  * Subject self-assessment
  * Independent evaluator assessment
  * Principal investigator assessment
  * Changes in RNA sequencing (from blood specimens)
  * Changes in MMP-1, Ang-2, VEGF and FGF (from blood specimens)

CONTACTS AND LOCATIONS:
Overall Officials: Lev Verkh, PhD, Study Director — Stemedica Cell Technologies, Inc.
Locations (2):
- United States (2):
  - eStudy Site, La Mesa, California
  - Naval Medical Center San Diego, San Diego, California